CLINICAL TRIAL: NCT01554826
Title: A Double - Blind, Randomized, - Controlled Clinical Trial With Inactivated Influenza Vaccine (Split Virion)(0.25ml Formulation for Pediatric Use)
Brief Title: Clinical Trial of the Inactivated Influenza Vaccine (0.25ml Formulation for Pediatric Use)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hualan Biological Engineering, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Hualanbio-influenza III-002
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-04

CONDITIONS: Influenza
Keywords: Pediatric influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza Split Vaccine (Experimental): 7.5μg HA/strain/0.25ml/syringe
  Interventions: Biological: Influenza Split Vaccine
- Inactivated Influenza Vaccine (Active Comparator): 7.5μg HA/strain/0.25ml/syringe
  Interventions: Biological: Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Split Vaccine — 0.25ml, two doses (540 subjects were randomly assigned to receive the first dose, among them, 515 subjects received a boost dose); two doses were assigned to be vaccinated 4 weeks apart
  Other Names: Hualan Biologicals
  Arms: Influenza Split Vaccine
Biological: Inactivated Influenza Vaccine — 0.25ml, two doses (270 subjects were randomly assigned to receive the first dose; among them, 263 subjects received a boost dose); two doses was administrated at 4 weeks apart
  Other Names: Vaxigrip, Shenzhen Aventis Pasteur Biological
  Arms: Inactivated Influenza Vaccine

SUMMARY:
The clinical trial was designed to evaluate the immunogenicity and safety against pediatric Inactivated influenza vaccine (Split Virion) (0.25ml formulation) of Hualan administered on infants age 6 months to 36 months.

DETAILED DESCRIPTION:
The clinical trial was designed randomized and double-blind. Participants included up to 810 persons (540 persons in test group and 270 persons in control group).

Healthy 6-36 months infants were selected, whose guardians were volunteers and had signed the informed consent. Subjects were selected according to the inclusion and exclusion criteria. Every subject accepted 30min's observation in the hospital after vaccination and received periodic follow-up till the fourth week after the boost vaccination.

Blood of subjects was collected at the third week after the boost vaccination for the analysis of the immunogenicity. During the test, the adverse reactions and detailed information were reported to the SFDA under the status of blinding every month. Unblinding was conducted after the completion of the follow-up of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Infants aging 6-36 months, their guardians understand and sign the informed consent
* Healthy infant by inquiring illness history, physical examination and clinical judgment and who complies with vaccination of this product
* Be able to comply with the requirement of clinical trial protocol
* Have no history of vaccination within the past 6 months and vaccination with other product within the latest 1 week
* Axillary temperature ≤37.0℃.

Exclusion Criteria:

1. Exclusion criteria for primary vaccination:

   * History of other vaccine or immunoglobulin inoculation within 2 weeks
   * History of eclampsia, epilepsy, encephalopathy and mental disease or family disease
   * History of vaccination allergy or allergy to drug and food (egg)
   * Known or suspected immunological function defects, including immunosuppressant therapy (radiotherapy, chemotherapy, corticosteroid hormone, antimetabolites, cytotoxic drug), genetic defects (favism), HIV infection or other reasons
   * Congenital malformation, maldevelopment or serious chronic disease (such as Down syndrome, diabetes, sickle cell anemia or neurologic disease)
   * Acute and chronic contagion, active infection (history of fever within the past 3 days (axillary temperature ≥38.0℃) or acute disease needing application of antibiotics or anti-virus treatment in the whole body)
   * Organic diseases such as liver, kidney, serious cardiovascular disease
   * Malignancy (tumor), serious asthma
   * Thrombopenia or other coagulopathy that may cause contraindication of intramuscular injection
   * Any condition resulting in the absence or removal the spleen
   * Hypertension (not including the higher blood pressure below 150mmHg and lower blood pressure below 100mmHg controlled by drug)
   * Participating in another clinical trial or any condition that, in the judgment of investigator, may affect trial assessment.
2. Exclusion criteria for a boost vaccination:

   * Any condition in the "Exclusion criteria" of the first injection after inclusion
   * Adverse reactions level 3 or above within 72 hours after first vaccination;
   * Serious adverse reactions having casual relationship with the first inoculation of test vaccine
   * Subjects are not willing to be inoculated any more and quit
   * Axillary temperature ≥37℃ before immunization
   * Reasons that can not conduct inoculation, in the judgment of investigators.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 810 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse reactions as a measure of safety study | 28 days after the vaccination
  Local reactions, systemic reactions, severity degree and AEFI correlation

SECONDARY OUTCOMES:
Observation of the immunogenicity | 28 days after the immunization
  HI antibody seroconversion ratios, protection ratios, GMTs and GMT increase folds

CONTACTS AND LOCATIONS:
Overall Officials: Feng-cai Zhu, M.D., Study Director — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Jiangsu Provincial Center for Disease Prevention and Control, Huaian, Jiangsu, China